CLINICAL TRIAL: NCT05894850
Title: Effect of the Automatic Surveillance System on Surveillance Rate of Colorectal Postpolypectomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EA-19-003-29
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Artificial Intelligence; Surveillance
Keywords: surveillance rate; automatic surveillance
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- With automatic surveillance system reminding through telephone and message (Experimental): Patients were reminded of the surveillance time by an automatic surveillance system after the endoscopic and pathological results were available and before the surveillance time through telephone and message.
  Interventions: Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS) reminds the patients through by telephone .; Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS) reminds the patients through message.
- With automatic surveillance system reminding through message (Experimental): Patients were reminded of the surveillance time by an automatic surveillance system after the endoscopic and pathological results were available and before the surveillance time through message.
  Interventions: Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS) reminds the patients through message.
- With manual reminder (Experimental): Patients were reminded of the surveillance time by manual reminder after the endoscopic and pathological results were available and before the surveillance time.
  Interventions: Other: Manually remind the patients
- Normal group (No Intervention): The patients in the control group were observed in the clinical natural state of surveillance without automatic surveillance system or manual reminder.

INTERVENTIONS:
Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS) reminds the patients through by telephone . — An automatic surveillance (AS) system to accurately identify post-polypectomy patients, assign surveillance intervals for different risks of patients and proactively follow up with patients at certain times. AI based automatic surveillance (AS) system (ENDOANGEL-AS) reminds patients by telephone.
  Arms: With automatic surveillance system reminding through telephone and message
Other: AI based automatic surveillance (AS) system (ENDOANGEL-AS) reminds the patients through message. — An automatic surveillance (AS) system to accurately identify post-polypectomy patients, assign surveillance intervals for different risks of patients and proactively follow up with patients at certain times. AI based automatic surveillance (AS) system (ENDOANGEL-AS) reminds patients through message.
  Arms: With automatic surveillance system reminding through message; With automatic surveillance system reminding through telephone and message
Other: Manually remind the patients — Medical staff remind patients manually .
  Arms: With manual reminder

SUMMARY:
In this study, we proposed a prospective study about the effect of the automatic surveillance system on surveillance rate of colorectal postpolypectomy patients. The enrolled patients were divided into group A with intelligent surveillance system reminding though telephone and message, group B with intelligent surveillance system reminding though message, group C with manual reminder, and group D with natural state. The surveillance among the four groups were compared.

DETAILED DESCRIPTION:
The adherence of doctors to published colorectal post-polypectomy surveillance guidelines varies greatly, and patient follow-up is critical but time-consuming. Previous studies we developed an automatic surveillance (AS) system to accurately identify post-polypectomy patients, assign surveillance intervals for different risks of patients and proactively follow up with patients in time. In this study, we proposed a prospective study about the effect of the automatic surveillance system on surveillance rate of colorectal postpolypectomy patients. The enrolled patients were divided into group A with intelligent surveillance system reminding though telephone and message, group B with intelligent surveillance system reminding though message, group C with manual reminder, and group D with natural state. The surveillance among the four groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older who undergo colonoscopy.

Exclusion Criteria:

* 1)No pathological result.
* 2) No or invalid contact information.
* 3) The surveillance interval cannot be determined according to the surveillance guidelines, including poor bowel preparation, colorectal cancer or suspicious malignance, surgery or colorectal ESD history, those who fail to complete colonoscopy due to unbearable, pathological indications of not polyps, hamartoma or lymphoma polyps, history of ulcerative colitis, and so on.
* 4) Has participated in other clinical trials, signed the informed consent form and is in the surveillance period of other clinical trials.
* 5) Have drug or alcohol abuse or psychological disorder in the past five years.
* 6）Pregnancy.
* 7）Not suitable for recruitment after investigator evaluation because of other high-risk conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1644 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
On-time Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with on-time surveillance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.

SECONDARY OUTCOMES:
Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with surveillance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.
Advance Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with surveillance in advance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.
Delayed Surveillance Rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with delayed surveillance, and the denominator is the number of all colorectal postpolypectomy patients requiring surveillance.
The accuracy of identifing post-polypectomy patients | 1 day At the time of enrollment
  The numerator is the number of patients correctly identified by automated surveillance system, and the denominator is the number of all enrolled colorectal postpolypectomy patients.
The accuracy of classifying risk levels | 1 day At the time of enrollment
  The numerator is the number of patients correctly classified by automated surveillance system, and the denominator is the number of all enrolled colorectal postpolypectomy patients.
The accuracy of assigning surveillance intervals | 1 day At the time of enrollment
  The numerator is the number of patients correctly assigned by automated surveillance system, and the denominator is the number of all enrolled colorectal postpolypectomy patients.
lesion progression rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion progression, and the denominator is the number of all surveillance colorectal postpolypectomy patients.
lesion persistence rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion persistence, and the denominator is the number of all surveillance colorectal postpolypectomy patients.
lesion regression rate | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with lesion regression, and the denominator is the number of all surveillance colorectal postpolypectomy patients.
The incidence rate of early colorectal cancer | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with early colorectal cancer in surveillance colonoscopy, and the denominator is the number of all surveillance colorectal postpolypectomy patients.
The incidence rate of colorectal cancer | From enrollment to study completion, assessed up to 3 years.
  The numerator is the number of patients with colorectal cancer in surveillance colonoscopy, and the denominator is the number of all surveillance colorectal postpolypectomy patients.

CONTACTS AND LOCATIONS:
Overall Officials: yuhonggang1969@163.com Yu, phD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No